CLINICAL TRIAL: NCT03806361
Title: Fat Grafts Supplemented With Adipose-derived Regenerative Cells for Soft Tissue Reconstruction in Children With Craniofacial Microsomia
Brief Title: Fat Grafts With Adipose-derived Regenerative Cells for Soft Tissue Reconstruction in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Daniela S Tanikawa, Principal investigator, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hospital Sirio Libanes
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Craniofacial Microsomia
MeSH Terms: conditions — Goldenhar Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, clinical trial with 2 parallel comparison groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will not know which treatment they will receive, outcome assessors will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With ADRC (Experimental): Supplementation of fat grafts with ADRC
  Interventions: Procedure: Fat grafts supplemented with ADRC
- Structural (Active Comparator): Structural fat grafting
  Interventions: Procedure: Structural fat grafting

INTERVENTIONS:
Procedure: Fat grafts supplemented with ADRC — Isolation of ADRC from fat aspirates and its use for supplementation of fat grafts.
  Arms: With ADRC
Procedure: Structural fat grafting — Fat grafts without supplementation of ADRC
  Arms: Structural

SUMMARY:
Although first reports of the clinical use of adipose-derived regenerative cells (ADRC) suggest that this approach may be feasible and effective for soft tissue augmentation, there is a lack of randomized, controlled clinical trials in the literature. Hence, this study aimed to investigate whether a novel protocol for isolation of ADRC and their use in combination with fat tissue improve the long-term retention of the grafts in paediatric patients with craniofacial microsomia.

DETAILED DESCRIPTION:
To overcome problems associated with fat grafting, such as unpredictable clinical results and a low rate of graft survival, many innovative efforts and refinements of surgical techniques have been reported. For example, condensation of living tissue and removal of unnecessary components have been performed by centrifugation, filtration or gravity sedimentation; external mechanical force has been used to expand the recipient tissue as well as the overlying skin envelope; and a recent experimental study has suggested that repeated local injections of erythropoietin might enhance retention of grafted fat.

Based on the finding that aspirated fat tissue contains a much smaller number of adipose-derived regenerative cells (ADRC) compared with intact tissue and that these cells play pivotal roles in the adipose tissue remodeling after lipoinjection, the supplementation of fat grafts with stromal vascular fraction isolated from adipose portion of liposuction aspirates has been proposed as a method to compensate its relative deficiency of ADRC.

In the literature, there are at least three experimental studies demonstrating that supplementation of adipose progenitor cells enhances the volume or weight of surviving adipose tissue, and first reports of the clinical use of ADRC suggest that this approach may be feasible and effective for soft tissue augmentation.

However, since these studies represent level of evidence IV, which correspond to the publication of case series, there is a lack of randomized, controlled clinical trials comparing this method to current standard techniques.

Hence, this study aimed to fill this gap by investigating whether a novel protocol for isolation of ADRC and their use in combination with fat tissue improve the long-term retention of the grafts in paediatric patients with craniofacial microsomia.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral craniofacial microsomia
* 10 to 18 years old
* Phenotype: (M0, M1 or M2) and (S1 or S2) according to the OMENS-Plus classification

Exclusion Criteria:

* Previous facial soft tissue surgery
* Absence of fat donor site

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Volumetric analysis of both hemifaces | Preoperative, 1 month postoperative, 3 months postoperative and 6 months postoperative
  Preoperative and 1, 3 and 6-months postoperative 3D-photogrammetry will be performed for volumetric measurements of both hemifaces using Vectra H1 software. Volumetric augmentation will be noticed for each patient by comparing the change between volumes of affected and unaffected hemifaces in the preoperative and 1, 3 and 6 months postoperative periods, which will be considered the retention volume. The percentage of fat graft survival will be determined as a ratio of the retention volume to the preoperative difference between volumes of affected and unaffected hemifaces.

SECONDARY OUTCOMES:
Number of viable cells | Intraoperative and immediate postoperative period
  Immediately after the surgical procedure the number of viable cells isolated before and after the supplementation of the grafts will be counted using the trypan blue dye exclusion assay in a Neubauer chamber using the light microscope Nikon Eclipse TS100 (Nikon Instruments Inc., NY, USA). Next, immunophenotype characterization of cell populations on passage 1 will be done by flow cytometric analysis with the anti-human antibodies CD29, CD31, CD45, CD90, CD73 and CD105 (Becton, Dickinson and Company, NJ, USA) in a Guava EasyCyte flow cytometer running the Guava Express Plus software (Guava Technologies Hayward, CA, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Municipal Infantil Menino Jesus, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No